CLINICAL TRIAL: NCT06335576
Title: Establishment of Serum Proteomics Subtypes of Gastric Cancer and Its Clinical
Brief Title: Establishment of Serum Proteomics Subtypes of Gastric Cancer and Its Clinical Application
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSGCproteomics
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric cancer patients receiving adjuvant chemotherapy
  Interventions: Other: This study is a single-arm and observational study with no intervention.

INTERVENTIONS:
Other: This study is a single-arm and observational study with no intervention. — This study is a single-arm and observational study with no intervention.

SUMMARY:
This study is a prospective, single-center, observational study aimed at detecting the status of serum protein profiles at key time points in gastric cancer patients receiving neoadjuvant therapy for advanced disease, and constructing a serum protein model for evaluating the efficacy of neoadjuvant therapy for gastric cancer. Subjects will receive neoadjuvant therapy (treatment regimen determined by the primary physician, limited to systemic therapy, with options including immune checkpoint inhibitor-based regimens and non-immune checkpoint inhibitor-based regimens). After four cycles of treatment, the efficacy will be assessed. Patients eligible for R0 resection will undergo D2 radical surgery regardless of tumor regression, while those ineligible for R0 resection will enter the palliative treatment phase (Note: Subjects are all patients who require neoadjuvant therapy even if they do not participate in this clinical study). Patients will receive regular follow-up evaluations for metastasis/recurrence and survival until tumor recurrence/progression or the last known date of patient survival (Note: Regular follow-up in this study follows the frequency of routine clinical follow-ups). The primary endpoint is progression-free survival (PFS), and the secondary endpoint is pathological response rate (based on Becker tumor regression grading, with residual tumor less than 50% considered effective preoperative treatment).

Peripheral venous blood samples will be collected before the start of neoadjuvant therapy (blood sampling point 1 - baseline) and before surgery after neoadjuvant therapy (blood sampling point 2 - post-treatment). Approximately 3 ml of blood will be collected each time, and about 1.5 ml of serum will be obtained after processing. Serum protein profiling will be conducted to assess the expression of protein profiles at these treatment time points.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 and ≤ 75 years old.
2. KPS score ≥ 80 points within 7 days prior to enrollment.
3. Histologically confirmed gastric adenocarcinoma at initial diagnosis.
4. Tumor located in the proximal stomach, including the gastroesophageal junction (defined as within 5cm proximal and distal to the cardia), gastric fundus, and upper body of the stomach.
5. Clinical staging based on endoscopic ultrasound or enhanced CT/MRI examination, staged as cT3~4aN+M0 (according to the 8th edition of AJCC TNM).
6. Presence of at least one evaluable lesion according to RECIST 1.1 criteria on abdominal CT/MRI examination.
7. Surgeon participating in this study determines that curative surgical resection is feasible.
8. Major organ function is able to tolerate neoadjuvant therapy.
9. No accompanying diseases that significantly reduce survival expectancy to < 5 years.
10. Willingness and ability to comply with the study protocol during the study period.
11. Provide written informed consent prior to entering the study, and the patient understands that they can withdraw from the study at any time without any loss.

Exclusion Criteria:

1. Patients with signs of distant metastasis or local unresectable factors.
2. Patients with imaging or endoscopic ultrasound suggesting T1 or T2 disease.
3. Patients who have received cytotoxic chemotherapy, radiotherapy, immunotherapy, or curative surgery for gastric cancer, excluding corticosteroids.
4. Patients who have experienced gastrointestinal bleeding within the two weeks prior to enrollment or are judged by the investigator to be at high risk of bleeding.
5. Patients with upper gastrointestinal obstruction, physiological dysfunction, or malabsorption syndrome that may affect oral drug absorption.
6. Patients who have received live vaccines within 4 weeks prior to enrollment. (Note: Seasonal influenza vaccines, which are usually inactivated vaccines, are allowed. Vaccines administered intranasally are live vaccines and are not allowed.)
7. Patients who have received immunotherapy (such as interleukins, interferons, thymosin, etc.) or any investigational treatment within 28 days prior to enrollment or within 5 half-lives (whichever is shorter, but at least 14 days).
8. Patients who have undergone major surgery within 28 days prior to enrollment, unless the surgery was minimally invasive (e.g., peripherally inserted central catheter [PICC] via peripheral venous puncture).
9. Uncontrolled systemic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in this study are gastric cancer patients receiving adjuvant chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
C-index | started 03-31-2024
  Effectiveness of the constructed serum protein model in predicting the efficacy of neoadjuvant chemotherapy for locally advanced gastric cancer (C-index)

SECONDARY OUTCOMES:
Sensitivity and specificity of model | started 03-31-2024
  Sensitivity and specificity of the constructed serum protein model in predicting the efficacy of neoadjuvant chemotherapy for locally advanced gastric cancer.